CLINICAL TRIAL: NCT01171417
Title: An Epidemiological Prospective Cohort Study to Describe Treatment Patterns of Fulvestrant And ExemeSTane in Postmenopausal Patients With Advanced HR+ Breast Cancer Under Real-life Conditions in GERmany
Brief Title: A Treatment With Fulvestrant and Exemestane in Postmenopausal Patients With Advanced Hormone Receptor-Positive (HR) + Breast Cancer
Acronym: ACT-FASTER:
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-ODE-FAS-2009/1; NIS-ODE-FAS-2009/1
Record Dates: First submitted 2010-06-23; First posted 2010-07-28 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Postmenopause; Breast Cancer
Keywords: Fulvestrant; Exemestane; postmenopausal patients; advanced HR+ breast cancer; Hormone Receptor positive; advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Cohort 1: 1st-line Faslodex 500 mg
- Cohort 2: 2nd-line Faslodex 500 mg
- Cohort 3: 3rd- line Faslodex 500 mg
- Cohort 4: patients on exemestane

SUMMARY:
For patients receiving Faslodex 500 mg, to compare the effectiveness in terms of Time to Progression (TTP) as a function of the line of treatment (i.e. 1st vs. 2nd vs. 3rd line). For all patients, to collect and explore real-life data on the epidemiology and management of Pseudomyxoma Peritonea (PMP) patients with HR+ advanced breast cancer (ABC) treated with Faslodex 500 mg or exemestane.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Female postmenopausal patient (or patient post-ovariectomy) and age ≥18 years Postmenopause ist defined as

  * Age ≥ 60 years and natural menopause with menses > 1year ago or
  * FSH and E2 levels in the postmenopausal range or
  * Patients who had bilateral ovariectomy (NCCN V.I. 2009)
* Histologically confirmed ER+ locally advanced or metastatic breast cancer
* Not eligible for curative therapy
* Prior treatment with tamoxifen
* Suitable to undergo endocrine treatment for ER+ ABC with SERD / sAI
* Patient is able to read and understand German

Exclusion Criteria:

* Known hypersensitivity to Faslodex or Exemestane or any compounds of the drugs
* Prior treatment with Faslodex 500 mg or Faslodex 250 mg*

  * for patients who receive treatment with Faslodex 500 mg within this observational study. Patients who are included in the exemestane arm may have received prior Faslodex treatment.
* Prior treatment with Exemestane for patients who receive treatment with Exemestane within this observational study
* Acutely life threatening disease
* Treatment with Faslodex 250 mg/month (previously approved dose)
* Prior palliative chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 660 patients in 140 sites in Germany. 100 specialists and 40 hospitals. Each site should enrol 4-20 patients
Sampling Method: Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effectiveness of Faslodex 500 mg in terms of time to progression (TTP) of disease. | Period from inclusion up to 9 months (average time period )
Disease management data | Period from inclusion up to 9 months (average time period )
  The analysis will be adjusted for the main prognostic factors, such as visceral metastases, age, receptor status etc

SECONDARY OUTCOMES:
Real-life data on patient outcomes by line of treatment (i.e. 1st vs. 2nd vs. 3rd line). | Every 3 months
  Including overall survival (OS), progression-free survival (PFS),time to progression (TTP), response rate (RR) and clinical benefit rate (CBR)
Real-life pharmacoeconomic data and use of health care resources. | Every 3 months
  According to lines of treatment and other patient related factors (such as age, co-morbidities etc.), including primary care visits, hospital stays and other resource
Health-related quality of life (HRQoL) in patients undergoing treatment with Faslodex 500 mg or exemestane. | Every 3 months
  Health-related quality of life will be assessed with a patient-based instrument (eg, EQ5D).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Maass, Prof. Dr. med., Principal Investigator — 52074 Aachen, Germany
Locations (92):
- Germany (92):
  - Research Site, Aachen
  - Research Site, Ahaus
  - Research Site, Amberg
  - Research Site, Aschaffenburg
  - Research Site, Aschersleben
  - Research Site, Bad Nauheim
  - Research Site, Bad Segeberg
  - Research Site, Bamberg
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bonn
  - Research Site, Böblingen
  - Research Site, Braunschweig
  - Research Site, Castrop-Rauxel
  - Research Site, Chemnitz
  - Research Site, Cologne
  - Research Site, Dachau
  - Research Site, Donauwurth
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Düsseldorf
  - Research Site, Eggenfelden
  - Research Site, Erfurt
  - Research Site, Eschweiler
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Euskirchen
  - Research Site, Frankfurt
  - Research Site, Frechen
  - Research Site, Freiburg im Breisgau
  - Research Site, Fürstenwalde
  - Research Site, Geesthacht
  - Research Site, Gera
  - Research Site, Goslar
  - Research Site, Göttingen
  - Research Site, Gröbenzell
  - Research Site, Hamburg
  - Research Site, Hanau
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Heidenheim
  - Research Site, Herdecke
  - Research Site, Hof
  - Research Site, Ilsede
  - Research Site, Ingolstadt
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kiel
  - Research Site, Landshut
  - Research Site, Langen
  - Research Site, Lehrte
  - Research Site, Ludwigsburg
  - Research Site, Lübeck
  - Research Site, Magdeburg
  - Research Site, Mayen
  - Research Site, Memmingen
  - Research Site, Mittweida
  - Research Site, Moers
  - Research Site, Mönchengladbach
  - Research Site, Mühlhausen
  - Research Site, München
  - Research Site, Münster
  - Research Site, Naunhof
  - Research Site, Nordhausen
  - Research Site, Nordhorn
  - Research Site, Nuremberg
  - Research Site, Oberhausen
  - Research Site, Offenbach
  - Research Site, Osnabrück
  - Research Site, Passau
  - Research Site, Plüderhausen
  - Research Site, Remagen
  - Research Site, Remscheid
  - Research Site, Rendsburg
  - Research Site, Rodewisch
  - Research Site, Rodgau
  - Research Site, Simmern
  - Research Site, Soest
  - Research Site, Stendal
  - Research Site, Stralsund
  - Research Site, Stuttgart
  - Research Site, Troisdorf
  - Research Site, Tübingen
  - Research Site, Villingen-Schwenningen
  - Research Site, Weiden
  - Research Site, Wetzlar
  - Research Site, Wiesbaden
  - Research Site, Worms
  - Research Site, Würselen
  - Research Site, Würzburg
  - Research Site, Zittau